CLINICAL TRIAL: NCT00360061
Title: Randomised Controlled Trial of Cognitive Behaviour Therapy: Efficacy and Acceptability for Adolescents With Type 1 Diabetes.
Brief Title: CBT in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bristol (Other)
Collaborators: Diabetes UK (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECCRA/2001; DUK grant BDA: RD01/0002114
Record Dates: First submitted 2006-08-01; First posted 2006-08-03 (Estimated); Last update posted 2006-08-03 (Estimated); Status verified 2001-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Adolescents; Cognitive Behaviour Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy

SUMMARY:
The effectiveness of cognitive behavioural therapy (CBT) for adolescents with type 1 diabetes will be tested. This structured, time-limited, problem-orientated therapy will be used to impact on psychosocial factors influencing diabetic control, with the patient and therapist working together on specific goals to develop adaptive strategies.

DETAILED DESCRIPTION:
Ninety 11-16 year olds with T1DM (duration >1 year), attending paediatric diabetes outpatient clinics based in 4 centres in South-West England, UK, will be recruited to a randomised controlled trial of one to one sessions of CBT versus non-directive supportive counselling. Participants will attend up to 6 sessions (weekly) with either a CBT therapist or a counsellor, with 2 further sessions at 6 and 12 months. Follow up will continue for 12 months post intervention. HbA1c is the primary outcome measure. Psychological measures will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Attendance at out-patients clinics at Bristol Royal Hospital for Children, Southmead Hospital in Bristol, Weston General Hospital, The Royal United Hospital in Bath, Gloucestershire Royal Hospital in Gloucester or the Musgrove Park branch of the Taunton and Somerset Hospital Aged 11-16 years old (inclusive) on the first day of the study Type 1 diabetes Duration at least 12 months on the first day of the study

Exclusion Criteria:

* chronic illnesses with dietary management implications (e.g. cystic fibrosis and coeliac disease) special educational needs (e.g. Down's syndrome) making the patient unable to co-operate with CBT in care of social services primary responsibility for care elsewhere English not spoken as a first language Known psychological/ psychiatric problems for which the patient has already been referred

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90
Dates: Start 2001-09; Study Completion 2005-06

PRIMARY OUTCOMES:
HBA1c

SECONDARY OUTCOMES:
Well Being Questionnaire, Children's Health locus of control,
Diabetes Quality of Life for Youths (modified from DCCT),
Self Efficacy for Diabetes Scale (modified version,),
Diabetes Family Behaviour Scale, Diabetes Readiness to Change Questionnaire,
Modified Health Care Climate Questionnaire (at baseline only).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Crowne, MD, Principal Investigator — UBHT; Ruth J Allen, PhD, Study Chair — University of Bristol
Locations (1):
- Bristol Royal Hospital for Children, Bristol, United Kingdom